CLINICAL TRIAL: NCT07237581
Title: Cognitive Behavioral Based Physical Therapy to Improve Functional Outcomes in Patients With Chronic Ankle Instability: a Pilot Randomized Control Trial
Brief Title: Cognitive Behavioral Based Physical Therapy for Patients With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Abbis Jaffri, Principal Investigator, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003479
Record Dates: First submitted 2023-06-21; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ankle Sprains; Chronic Ankle Instability
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: investigators involved in participant screening, outcome measures, and intervention administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBPT/HEP Group (Experimental): Participants receive six sessions (45 minutes each) of a CBPT program, consisting of behavioral self-management, problem solving, cognitive restructuring, and relaxation training. Participants also receive 3 weeks of a home exercise physical therapy program, consisting of flexibility, foot and ankle strengthening, and balance exercises.
  Interventions: Behavioral: CBPT/HEP
- HEP Only Group (Active Comparator): Participants receive 3 weeks of a home exercise physical therapy program, consisting of flexibility, foot and ankle strengthening, and balance exercises.
  Interventions: Behavioral: HEP Only

INTERVENTIONS:
Behavioral: CBPT/HEP — 6 sessions of CBPT program and 3 weeks HEP
  Arms: CBPT/HEP Group
Behavioral: HEP Only — 3 weeks HEP
  Arms: HEP Only Group

SUMMARY:
The purpose of this study is to investigate the feasibility of a psychologically informed physical therapy intervention in individuals with Chronic Ankle Instability.

DETAILED DESCRIPTION:
This project will target the psychological impairments in addition to pathomechanical and motor behavior impairment in individuals with Chronic Ankle Instability, using a cognitive behavioral based physical therapy approach. All participants will first complete a baseline assessment, then will be randomly assigned to treatment groups (CBPT/home exercise program (HEP) or HEP only) using a random number generator by an investigator not involved in participant screening, outcome measures, or intervention administration. Individuals in the CBPT/HEP group will participate in six sessions of 45 minutes each for three weeks (two sessions a week). After three weeks, a post-assessment will be completed for both groups.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one ankle sprain (initial sprain at least 1 year prior to participation)
* Reported foot and ankle ability measure-sports scale (FAAM-sport) <85, identification of functional ankle instability (IdFAI) >10

Exclusion Criteria:

* History of other lower extremity fracture or surgery
* Ankle sprain within the past 6-weeks
* Any conditions known to affect balance
* Pregnancy
* Any neurological or psychological problems
* Individuals already participating in rehabilitation

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Number of Prescribed Sessions Attended per Subject | 3 weeks
  At least 85% of subjects must complete follow-up testing. A subject who attends post-intervention visit at 3 weeks has completed the follow-up testing.
Percentage of Subjects Completing All Prescribed Sessions Within 3 Weeks | 3 weeks
  At least 80% of subjects must attend all the sessions prescribed. Attendance means the subject has showed up and completed the tasks for the session.
Number of Intervention-Related Serious Adverse Events Per Group Within 3 Weeks | 3 weeks
  Adverse events are recorded as unfavorable events in which a subject has unintentional and abnormal signs or symptoms temporarily associated with participation in the intervention. The number of adverse events in the intervention group should be similar to that of the control group and will not exceed three serious adverse events related to the intervention.
Change from baseline kinesiophobia at 3 weeks (post-intervention) | 3 weeks
  The Tampa Scale of Kinesiophobia (11-question version), which uses a 4-point Likert scale, will be used to assess fear of movement. Individual item scores range from 1-4. Total score is the sum of all scores. Minimum possible total score is 11 and maximum possible total score is 44. Higher scores indicate a worse outcome or greater fear of movement.
Change from baseline self-efficacy at 3 weeks (post-intervention) | 3 weeks
  Self-efficacy will be assessed using the 17-item self-efficacy questionnaire. 17 statements of physical activity are scored from 0-100% according to subject's perceived ability to carry out the tasks in the statement. Total score is the average of all scores. Higher scores represent a better outcome or greater self-efficacy.
Change from baseline health related quality of life at 3 weeks (post-intervention) | 3 weeks
  Health related quality of life will be assessed using the Disablement in the Physically Active Scale. Individual scores range from 0-4. Total scores are calculated as a sum of individual scores. 2 sub-scales (physical summary component and mental summary component) are calculated along with a total score. Physical summary component scores range from 0-48. Mental summary component scores range from 0-16. Total scores range from 0-64. Higher scores represent worse outcome or worse health related quality of life.
Change from baseline physical activity at 3 weeks (post-intervention) | 3 weeks
  Physical activity will be measured by daily steps recorded using Actigraph activity monitor watches.
Change from baseline foot and ankle range of motion at 3 weeks (post-intervention) | 3 weeks
  Foot and ankle range of motion will be measured using clinical goniometry techniques and recorded in the unit of degrees.
Change from baseline dynamic balance at 3 weeks (post-intervention) | 3 weeks
  Dynamic balance will be measured using a modified Star Excursion Balance Test and reported as a relative distance (%).

SECONDARY OUTCOMES:
Change from baseline center of force anterior-posterior excursion balance (cm) | 3 weeks
  Measurements will be taken using a Tekscan pressure mat in a single-leg balance test and recorded in units of cm.
Change from baseline center of force left-right excursion balance (cm) | 3 weeks
  Measurements will be taken using a Tekscan pressure mat in a single-leg balance test and recorded in units of cm.
Change from baseline foot and ankle muscle strength (Newtons) | 3 weeks
  Foot and ankle muscle strength will be measured using hand held dynamometry and reported in units of Newtons.
Change from baseline center of force total area (cm^2) | 3 weeks
  Center of force will be measured using a Tekscan pressure mat in a single-leg balance test and recorded in units of cm^2.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Science Research Lab, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No